CLINICAL TRIAL: NCT01116635
Title: Phase I/II Study Examining Pharmacokinetics, Adverse Events, and Surgically Resected Histopathological Response Utilizing a Dose Escalation Model of Doxorubicin Loaded Drug Eluting Superabsorbent Polymer Microspheres in Surgically Resectable Hepatocellular Carcinoma in Humans
Brief Title: Clinical Study Examining the Safety and Efficacy of Doxorubicin Drug Eluting Microspheres Transarterial Embolization in the Setting of Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H08-02833
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: chemoembolization; drug eluting microsphere; hepato; embolotherapy; downstage
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin; Embolization, Therapeutic; Chemoembolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 50mg dose loading per vial of doxorubicin (Experimental)
  Interventions: Drug: doxorubicin, superabsorbent polymer microspheres, embolotherapy
- 75mg dose loading per vial of doxorubicin (Experimental)
  Interventions: Drug: doxorubicin, superabsorbent polymer microspheres, embolotherapy

INTERVENTIONS:
Drug: doxorubicin, superabsorbent polymer microspheres, embolotherapy — varying doses of doxorubicin loaded onto SAP during embolization procedure. Pharmacokinetic analysis of elution profile through serum concentrations over 1 month period embolization of surgically resectable HCC with superabsorbent polymer microspheres loaded with doxorubicin from a single treatment. Phase I will follow a modified Fibonacci sequence (with pharmacokinetic analysis of serum doxorubicin) to determine mean tolerated dose (MTD), severe adverse reaction (SAE) and dose limiting toxicities (DLT) when microspheres are loaded with 25mg, 50mg, or 75mg of doxorubicin. Phase II will continue enrollment with the two highest tolerated doses. At least one month after treatment, all patients will undergo imaging and surgical resection of reference tumor, with assessment of degree of necrosis, microsphere distribution, and correlation with concentration of doxorubicin loaded onto microsphere.
  Other Names: chemoembolization; drug eluting bead; drug eluting microsphere; superabsorbent microsphere; radioembolization; bland embolization

SUMMARY:
The study is designed to determine whether loading doxorubicin (a type of chemotherapy), when loaded onto a drug eluting microsphere will result in increased destruction of a tumor. The study will treat patients with surgically resectable liver cancers with varying doses of doxorubicin loaded into microspheres, with a close review of any side effects and chemotherapy concentrations in the bloodstream. The tumors will be surgically removed after at least 1 month, to determine how much the tumor has shrunk, and the amount of tumor destroyed. It is hoped that the study results will determine if this treatment has a role in controlling tumor growth prior to surgical removal.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with surgically resectable hepatocellular carcinoma (HCC)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Histopathological correlation with surgically resected tumor

SECONDARY OUTCOMES:
Dose limiting toxicities
serum doxorubicin release patter
maximum tolerated dose

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chung, MD, Study Director — University of British Columbia; Jo-Ann Ford, RN, Study Director — University of British Columbia; Sharlene Gill, MD, Study Director — University of British Columbia; Stephen Ho, MD, Study Director — University of British Columbia; David Owen, MD, Study Director — University of British Columbia; Charles Scudamore, MD, Study Director — University of British Columbia; Ellen Wasan, PhD, Study Director — University of British Columbia; Alan Weiss, MD, Study Director — University of British Columbia; Eric Yoshida, MD, Study Director — University of British Columbia; Sigfried Erb, MD, Study Director — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Klass D, Owen D, Buczkowski A, Chung SW, Scudamore CH, Weiss AA, Yoshida EM, Ford JA, Ho S, Liu DM. The effect of doxorubicin loading on response and toxicity with drug-eluting embolization in resectable hepatoma: a dose escalation study. Anticancer Res. 2014 Jul;34(7):3597-606. PMID 24982375